CLINICAL TRIAL: NCT02365766
Title: Phase Ib/II Study of Neoadjuvant Pembrolizumab With Gemcitabine-Cisplatin (Cisplatin-Eligible) or Gemcitabine (Cisplatin-Ineligible) in Subjects With T2-4aN0M0 Urothelial Cancer: HCRN GU14-188
Brief Title: Neoadjuvant Pembrolizumab in Combination With Gemcitabine Therapy in Cis-eligible/Ineligible UC Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jason R. Brown (Other)
Collaborators: Hoosier Cancer Research Network (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Jason R. Brown, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU14-188
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
Keywords: MK-3475; Gemcitabine; Cisplatin; Pembrolizumab; Neoadjuvant Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — pembrolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A - Phase 1b Dose Finding Cohort: (Experimental): Cisplatin-eligible subjects will receive pembrolizumab at starting dose of 200mg (dose level 0), and/or 120mg (dose level -1) in combination with gemcitabine and cisplatin. The MTD will be the highest pembrolizumab dose level in combination with gemcitabine/cisplatin every 21 days, repeated for 4 cycles. (Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days). Once the MTD is established, this portion of the study will close and the phase II will open to cohorts I and II at the recommended phase II dose (RP2D).
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin
- Arm B - Phase II Cohort I: (Experimental): Cisplatin-eligible subjects receive gemcitabine/cisplatin every 21 days, repeated for 4 cycles. (Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days) . Pembrolizumab at RP2D is given every 21 days for 5 doses starting C1D8. Note: the last dose of pembrolizumab falls on what would be day 8 of a 5th 'chemo' cycle, however gemcitabine/cisplatin is NOT GIVEN. Subjects will then have consolidative surgery to remove their primary tumor within 2-7 weeks after their last dose of neoadjuvant therapy.
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin; Procedure: Consolidative Surgery
- Arm C - Phase II Cohort II: (Experimental): Cisplatin-ineligible subjects receive gemcitabine every week every 28 days for 3 cycles. Pembrolizumab at RP2D is given every 21 days for 5 doses starting C1D8. NOTE: due to the timing of gemcitabine cycles every 4 weeks, and every 3-week dosing of pembrolizumab, there are two doses of pembrolizumab given during cycle 2: D1 and D22. Additionally, the last dose of pembrolizumab falls on what would be D8 of a 4th 'chemo' cycle; however gemcitabine is NOT GIVEN. Subjects will then have consolidative surgery to remove their primary tumor within 2-7 weeks after their last dose of neoadjuvant therapy.
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Procedure: Consolidative Surgery

INTERVENTIONS:
Drug: Pembrolizumab — In this dose-finding cohort, pembrolizumab (MK-3475) will be administered (cisplatin-eligible patients only) at starting dose 200mg IV every 21 days for 4 cycles to determine RP2D. Once MTD is established in phase Ib, pembrolizumab will be administered on phase II cohorts I and II at RP2D every 21 days for 5 cycles.
  Other Names: MK-3475
Drug: Gemcitabine — For cisplatin-eligible patients on phase Ib and phase II cohort 1, gemcitabine 1000mg/m2 IV, D1 and D8 every 21 days for 4 cycles. For cisplatin-ineligible patients on phase II cohort II, gemcitabine 1000mg/m2 will be administered D1, D8 and D15 every 28 days for 3 cycles.
  Other Names: Gemzar
Drug: Cisplatin — For cisplatin-eligible patients, cisplatin 70mg/m2 IV will be administered D1 every 21 days for 4 cycles.
  Other Names: Platinol
  Arms: Arm A - Phase 1b Dose Finding Cohort:; Arm B - Phase II Cohort I:
Procedure: Consolidative Surgery — Following completion of treatment, subjects will then have surgery to remove their primary tumor within 2-7 weeks after their last dose of neoadjuvant therapy.
  Arms: Arm B - Phase II Cohort I:; Arm C - Phase II Cohort II:

SUMMARY:
This is a pre-surgical study involving subjects with muscle invasive bladder cancer, or urothelial cancer, who are candidates for neoadjuvant therapy. It is is a two-part trial with a one-arm phase Ib portion followed by a two-arm phase II portion. The study treatment is stratified into two cohorts based on cisplatin eligibility.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

INVESTIGATIONAL TREATMENT:

Phase Ib Dose-Finding Cohort I Cisplatin-Eligible:

Phase Ib is a 3+3 design for the cisplatin-eligible group only. Cisplatin-eligible subjects receive: gemcitabine 1000mg/m2 IV D1 and D8 every 21 days repeated for 4 cycles; cisplatin 70mg/m2 IV D1 and D8 every 21 days, repeated for 4 cycles. (Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days). Pembrolizumab will be given every 3 weeks for 5 doses, with a starting dose of 200 mg. NOTE: the last dose of pembrolizumab falls on what would be D8 of a 5th 'chemo' cycle, however gemcitabine/cisplatin is NOT GIVEN.

Phase II Arm A: Cohort I Cisplatin-Eligible:

Cisplatin-eligible subjects receive: gemcitabine 1000mg/m2 IV D1 and D8 every 21 days repeated for 4 cycles; cisplatin 70mg/m2 IV D1 and D8 every 21 days, repeated for 4 cycles. (Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days). Pembrolizumab at recommended phase II dose (RP2D) is given every 3 weeks for 5 doses starting with C1D8. NOTE: the last dose of pembrolizumab falls on what would be day 8 of a 5th 'chemo' cycle, however gemcitabine/cisplatin is NOT GIVEN. Cohort I treatment with gemcitabine and cisplatin will continue for a maximum of 4 cycles (cycle = 21days).

Phase II Arm B: Cohort II:

Cisplatin-ineligible subjects receive gemcitabine 1000mg/m2 IV D1, D8 and D15 every 28 days, repeated for 3 cycles. Pembrolizumab at RP2D is given every 3 weeks for 5 doses starting with C1D8. NOTE: due to the timing of gemcitabine cycles every 4 weeks, and every three week dosing of pembrolizumab, there are two doses of pembrolizumab given during cycle 2: D1 and D22. Additionally, the last dose of pembrolizumab falls on what would be D8 of a 4th 'chemo' cycle; however gemcitabine is NOT GIVEN. Cohort II treatment with gemcitabine will continue for a maximum of 3 cycles (cycle = 28 days)

Subjects will then have surgery to remove their primary tumor within 2-7 weeks after their last dose of neoadjuvant therapy.

Eastern Cooperative Oncology Group (ECOC) performance status: 0-1 for cisplatin-eligible subjects; 0-2 for cisplatin-ineligible subjects.

Demonstrate adequate organ function as defined by the following laboratory values at study entry. All screening labs should be performed within 28 days of C1D1.

Hematopoetic:

* Absolute neutrophil count (ANC) ≥1,500 /mcL
* Absolute lymphocyte count ≥350 mcL
* Platelets ≥100,000 / mcL
* Hemoglobin ≥9 g/dL or ≥5.6 mmol/L

Renal:

* Measured or calculated creatinine clearance ≥30 mL/min

Hepatic:

* Serum total bilirubin ≤ 1.25 X ULN OR ≤ 2.5 x ULN for subjects with Gilbert's disease
* Aspartate aminotransferase (AST, SGOT) and alanine aminotransferase (ALT, SGPT) ≤ 2 X ULN

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy and as long as PT or PTT is within therapeutic range of intended use of anticoagulants

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Over 18 years of age on day of signing informed consent.
* ECOG PS ≤ 2; please see protocol for specific details regarding ECOG PS for each cohort.
* Have histologically confirmed muscle invasive disease of the urinary bladder. For subjects who have tumors limited to the upper tract including renal pelvis or ureters, muscle invasive disease does not need to be pathologically proven, and a CT urogram must be performed (MRI is not acceptable to meet this criterion). To be eligible, subjects with upper tract tumors of the renal pelvis and ureter(s) must meet a high risk assessment defined as: tumor ≥ 1cm and/or hydronephrosis and/or high grade pathology and/or multifocal disease, where a radical NU approach to treat localized disease is warranted.
* Histology must be urothelial carcinoma (transitional cell carcinoma) or urothelial carcinoma with mixed histology/features.
* Clinical stage cT2-4aN0M0. Please see exclusion criteria for acceptable N0 determination/lymph node size.
* Have a surgical evaluation that documents the plan for multimodality therapy with a consolidative radical cystectomy or nephroureterectomy.

NOTE on surgical intent: Criteria for acceptable surgical risk are not defined and per treating urologist. Minimum guidance on surgical intent includes subjects who do not have significant cardiovascular disease such as NHYA class III or IV heart failure, unstable arrhythmias or angina, active CAD, and/or EF<25%. Specific diagnostic testing to determine surgical intent is not required and per treating urologist or oncologist discretion.

* Having an archived tumor block available to submit 11 unstained slides for PD-L1 expression, basal and luminal subtype analysis is MANDATORY for subjects with bladder cancer (optional for those with tumors limited to the upper tract if sufficient tissue is not available). If slides are not available, a biopsy is strongly encouraged to obtain tissue for submission (See Study Procedures Manual for collection, labeling and shipping instructions).
* Subjects on full dose anticoagulants must be on a stable regimen of warfarin or low molecular weight heparin (LMWH) for at least two weeks.
* Demonstrate adequate organ function as defined below: All screening labs should be performed within 28 days of study registration.
* System

  * Hematological

    * Absolute neutrophil count (ANC): ≥1500 / mcL
    * Absolute lymphocyte count: ≥350 mcL
    * Platelets: ≥100,000/mcL
    * Hemoglobin: ≥9 g/dL or ≥5.6 mmol/L
  * Renal

    ---Measured or calculated creatinine clearance: ≥30 mL/min
  * Hepatic

    * Serum total bilirubin: ≤1.25 X ULN OR ≤2.5xULN for subjects with Gilbert's disease
    * AST(SGOT) and ALT(SGPT): ≤2 X ULN
  * Coagulation

    * International Normalized Ratio (INR) or Prothrombin Time (PT): ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
    * Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN unless subject is receiving anticoagulant therapy and as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to study registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required.
* Female subjects of childbearing potential must be willing to use 2 methods of birth control, be surgically sterile, or abstain from heterosexual intercourse for the course of the study and through 120 days after the last dose of study medication. NOTE: Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects must agree to use a barrier method of male contraception starting with the first dose of study therapy and through 120 days after the last dose of study therapy.

COHORT I - CISPLATIN-ELIGIBLE:

In addition to the inclusion criteria listed above, Cohort I subjects must satisfy all of the following criteria:

* Glomerular filtration rate (GFR) or creatinine clearance (Ccr) ≥ 50 mL/min. (24 hour urine preferred). The cisplatin dose will be split over two days for values between 50-59 mL/min
* ECOG PS 0, 1 (and not 2)
* Hearing impaired ≤ grade 1 (may or may not be enrolled in a monitoring program)
* Peripheral neuropathy ≤grade 1

COHORT II - CISPLATIN-INELIGIBLE:

In addition to the inclusion criteria listed above, Cohort II subjects must also meet any ONE of the following criteria:

* GFR or Ccr: 30-49 (24 hour urine preferred).
* ECOG PS 2
* Hearing impaired ≥grade 2 as assessed by treating physician (may or may not be enrolled in a monitoring program).
* Peripheral neuropathy of Grade 2-4

Exclusion Criteria:

Subjects may not have any of the following:

* A non-surgical approach recommended by the treating urologist due to any reason. Criteria for surgical intent are not defined and, rather, suitability is determined and documented by the subject's treating urologist. Minimum guidance on surgical intent includes subjects who do not have significant cardiovascular disease such as NHYA class III or IV heart failure, unstable arrhythmias or angina, active CAD, and/or EF<25%. Specific cardiopulmonary diagnostic testing to determine surgical intent is not required and per treating urologist or oncologist discretion.
* Has abdomino-pelvic short axis lymph node of ≥15mm without biopsy. NOTE: A subject with a staging biopsy proving a non-neoplastic process/N0 will meet inclusion.
* Subjects with disease that is limited to the upper tract urothelial cancer and is considered low risk defined as: unifocal disease and tumor size <1cm, and low grade cytology, and without an invasive aspect on CT-urography.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 28 days prior to study registration.
* Has a diagnosis of immunodeficiency or received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration. Subjects on steroids for physiologic replacement due to a non-cancer related cause would not be excluded.
* Has had a prior monoclonal antibody ≤ 28 days prior to study registration or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 28 days earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy for urothelial carcinoma.
* Has a known additional malignancy that is progressing or required treatment ≤ 48 months of study registration. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer that has undergone potentially curative therapy, stable (as defined by PSA change, checked within 30 days) and untreated very low-risk or low-risk prostate cancer defined by current NCCN guidelines.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Brain imaging is not required and per discretion of treating physician.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
* Has known evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received therapy with hematopoietic growth factor such as G-CSF or GM-CSF in the 14 days prior to registration.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to the first dose of trial treatment. NOTE: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccines. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason R. Brown, M.D.,PhD, Study Chair — Hoosier Cancer Research Network
Locations (9):
- United States (9):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Care, Indianapolis, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - Washington University: Siteman Cancer Center, St Louis, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Thomas Jefferson University: Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants in Phase 1b received same dose (Pembrolizumab 200 mg).
Groups:
- Phase 1b Cohort I: Cisplatin-eligible - Pembrolizumab 200 mg: Arm A: Cisplatin-eligible subjects were received pembrolizumab at starting dose of 200mg (dose level 0) in combination with gemcitabine and cisplatin. Once the MTD is established, this portion of the study will close and the phase II will open to cohorts I and II at the recommended phase II dose (RP2D).
  Pembrolizumab: In this dose-finding cohort, pembrolizumab (MK-3475) were administered (cisplatin-eligible patients only) at starting dose 200mg IV every 21 days for 4 cycles to determine RP2D. Once MTD is established in phase Ib, pembrolizumab will be administered on phase II cohorts I and II at RP2D every 21 days for 5 cycles.
  Gemcitabine: For cisplatin-eligible patients on phase Ib, gemcitabine 1000mg/m2 IV, D1 and D8 every 21 days for 4 cycles.
  Cisplatin: For cisplatin-eligible patients, cisplatin 70mg/m2 IV will be administered D1 every 21 days for 4 cycles.
- Phase II Cohort I: Cisplatin-eligible- Pembrolizumab 200 mg: Arm B: Cisplatin-eligible subjects receive gemcitabine/cisplatin every 21 days, repeated for 4 cycles. (Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days) . Pembrolizumab at RP2D is given every 21 days for 5 doses starting C1D8. Note: the last dose of pembrolizumab falls on what would be day 8 of a 5th 'chemo' cycle, however gemcitabine/cisplatin is NOT GIVEN. Subjects will then have consolidative surgery to remove their primary tumor within 2-7 weeks after their last dose of neoadjuvant therapy.
  Pembrolizumab: Once MTD is established in phase Ib, pembrolizumab will be administered on phase II cohorts I and II at RP2D every 21 days for 5 cycles.
  Gemcitabine: For cisplatin-eligible patients on phase II cohort 1, gemcitabine 1000mg/m2 IV, D1 and D8 every 21 days for 4 cycles.
  Cisplatin: For cisplatin-eligible patients, cisplatin 70mg/m2 IV will be administered D1 every 21 days for 4 cycles.
- Phase II Cohort II: Cisplatin-ineligible -Pembrolizumab 200 mg: Arm C: Cisplatin-ineligible subjects receive gemcitabine every week every 28 days for 3 cycles. Pembrolizumab at RP2D is given every 21 days for 5 doses starting C1D8. NOTE: due to the timing of gemcitabine cycles every 4 weeks, and every 3-week dosing of pembrolizumab, there are two doses of pembrolizumab given during cycle 2: D1 and D22. Additionally, the last dose of pembrolizumab falls on what would be D8 of a 4th 'chemo' cycle; however gemcitabine is NOT GIVEN. Subjects will then have consolidative surgery to remove their primary tumor within 2-7 weeks after their last dose of neoadjuvant therapy.
  Pembrolizumab: Once MTD is established in phase Ib, pembrolizumab will be administered on phase II cohorts I and II at RP2D every 21 days for 5 cycles.
  Gemcitabine: For cisplatin-ineligible patients on phase II cohort II, gemcitabine 1000mg/m2 will be administered D1, D8 and D15 every 28 days for 3 cycles.
Period: Overall Study
Arm/Group | Phase 1b Cohort I: Cisplatin-eligible - Pembrolizumab 200 mg | Phase II Cohort I: Cisplatin-eligible- Pembrolizumab 200 mg | Phase II Cohort II: Cisplatin-ineligible -Pembrolizumab 200 mg
Started | 6 | 37 | 40
Completed | 6 | 37 | 38
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Eligibility Criteria Not Met | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b Cohort I: Cisplatin-eligible - Pembrolizumab 200 mg | Phase II Cohort I: Cisplatin-eligible- Pembrolizumab 200 mg | Phase II Cohort II: Cisplatin-ineligible -Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 6 | 37 | 38 | 81
Age, Continuous [Median (Full Range); unit: years] | 66 [58 to 74] | 63 [42 to 77] | 73 [58 to 83] | 68 [42 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 10 | 11 | 22
  Male | 5 | 27 | 27 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 35 | 36 | 77
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 3 | 9
  White | 5 | 31 | 35 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 37 | 38 | 81
ECOG performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    ECOG = 0 | 6 | 26 | 22 | 54
    ECOG = 1 | 0 | 11 | 12 | 23
    ECOG = 2 | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Safety of Pembrolizumab in Combination With Gemcitabine-Cisplatin
Description: Number of patients with experienced Dose-Limiting Toxicities (DLTs) will be monitored as a safety and tolerability of pembrolizumab in combination with gemcitabine and cisplatin . The Pembrolizumab DLT is defined as a drug-related adverse events (AEs) per Common Terminology Criteria for Adverse Events (CTCAE) V4 criteria that occurs in the first 4 weeks of treatment of pembrolizumab (C1D8 - C2D14) and meets the DLT definition per protocol.
Time Frame: Up to 4 weeks
Population: All participants in Phase 1b received same dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort I: Cisplatin-eligible - Pembrolizumab 200 mg
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Rate of Pathologic Muscle Invasive Response (PaIR)
Description: Pathologic muscle invasion response (PaIR), or ≤ypT1N0M0, rate is assessed from the consolidative surgery (radical cystectomy (RC) / nephroureterectomy (NU) - lymph node dissection (LND)) specimen.
Time Frame: Within 2-7 weeks post last dose of pembrolizumab (up to 6 months)
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint PaIR Rate was defined as all Cisplatin-eligible treated at the MTD, which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2 + cisplatin 70mg/m2; and all Cisplatin-ineligible treated at the MTD which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2.
  38 out of 43 Cisplatin eligible patients and 33 out of 38 Cisplatin ineligible patients had data of pathological response.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg: Cisplatin eligible (receive treatment in Phase Ib and II) : Cisplatin eligible subjects receive gemcitabine/cisplatin every 3 weeks, repeated for 4 cycles. Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days.
  Pembrolizumab is given every 3 weeks for 5 doses starting with Cycle 1 Day 8 (C1D8).
  NOTE: the last dose of pembrolizumab falls on what would be day 8 of a 5th 'chemo' cycle, however gemcitabine/cisplatin is NOT GIVEN
- Cohort II: Cisplatin Ineligible - Pembrolizumab 200 mg: Cisplatin ineligible (receive treatment in Phase II only) : Cisplatin ineligible subjects receive gemcitabine every week (weekly) for three consecutive weeks, repeated every 28 days for 3 cycles. Pembrolizumab is given every 3 weeks for 5 doses starting with Cycle 1 Day 8 (C1D8). NOTE: due to the timing of gemcitabine cycles every 4 weeks, and every three week dosing of pembrolizumab, there are two doses of pembrolizumab given during cycle 2: days 1 and 22. Additionally, the last dose of pembrolizumab falls on what would be day 8 of a 4th 'chemo' cycle; however gemcitabine is NOT GIVEN.
Arm/Group | Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg | Cohort II: Cisplatin Ineligible - Pembrolizumab 200 mg
Number analyzed (Participants) | 38 | 33
Percentage of participants | 61 [46 to 74] | 51.5 [35 to 68]

3. Secondary Outcome: Relapse-Free Survival (RFS) at 18 Months
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Relapse-Free Survival is defined by the date of randomization until the criteria for disease progression is met as defined by RECIST 1.1 or death occurs.
Time Frame: 18 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Relapse-Free Survival was defined as all Cisplatin-eligible patients treated at the MTD, which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2 + cisplatin 70mg/m2; and all Cisplatin-ineligible patients treated at the MTD which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2.
  37 out of 38 Cisplatin ineligible patients were evaluable for RFS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort II: Cisplatin Ineligible - Pembrolizumab 200 mg: Cisplatin ineligible (receive treatment in Phase II only): Cisplatin ineligible subjects receive gemcitabine every week (weekly) for three consecutive weeks, repeated every 28 days for 3 cycles. Pembrolizumab is given every 3 weeks for 5 doses starting with Cycle 1 Day 8 (C1D8). NOTE: due to the timing of gemcitabine cycles every 4 weeks, and every three week dosing of pembrolizumab, there are two doses of pembrolizumab given during cycle 2: days 1 and 22. Additionally, the last dose of pembrolizumab falls on what would be day 8 of a 4th 'chemo' cycle; however gemcitabine is NOT GIVEN.
Arm/Group | Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg | Cohort II: Cisplatin Ineligible - Pembrolizumab 200 mg
Number analyzed (Participants) | 43 | 37
Percentage of participants | 83 [67 to 91] | 57.4 [40 to 72]

4. Secondary Outcome: Overall Survival (OS) at 5 Years
Description: Determine the Overall survival at 5 years. OS is defined by the date of randomization to date of death from any cause.
Time Frame: 5 years
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Overall Survival was defined as all Cisplatin-eligible patients treated at the MTD, which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2 + cisplatin 70mg/m2; and all Cisplatin-ineligible patients treated at the MTD which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg | Cohort II: Cisplatin Ineligible - Pembrolizumab 200 mg
Number analyzed (Participants) | 43 | 38
Percentage of participants | 71.9 [55 to 83] | 56.6 [39 to 71]

5. Secondary Outcome: Radical Cystectomy (RC) Rate
Description: To compare the radical cystectomy (RC) rates in subjects who are cisplatin-eligible with those who are cisplatin-ineligible.
Time Frame: Within 2-7 weeks post last dose of pembrolizumab (up to 6 months)
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Radical Cystectomy Rate was defined as all Cisplatin-eligible patients treated at the MTD, which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2 + cisplatin 70mg/m2; and all Cisplatin-ineligible patients treated at the MTD which was determined to be pembrolizumab 200 mg + gemcitabine 1000mg/m2.
  37 out of 38 Cisplatin ineligible patients were evaluable for Radical Cystectomy Rate.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg: Cisplatin eligible (receive treatment in Phase Ib and II): Cisplatin eligible subjects receive gemcitabine/cisplatin every 3 weeks, repeated for 4 cycles. Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days.
  Pembrolizumab is given every 3 weeks for 5 doses starting with Cycle 1 Day 8 (C1D8).
  NOTE: the last dose of pembrolizumab falls on what would be day 8 of a 5th 'chemo' cycle, however gemcitabine/cisplatin is NOT GIVEN
Arm/Group | Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg | Cohort II: Cisplatin Ineligible - Pembrolizumab 200 mg
Number analyzed (Participants) | 43 | 37
Percentage of participants | 86 [73 to 93] | 89 [76 to 96]

ADVERSE EVENTS:
Time Frame: Up to a maximum of 5 years
Groups:
- Phase 1b Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg: Cisplatin-eligible subjects were received pembrolizumab at starting dose of 200mg (dose level 0) in combination with gemcitabine and cisplatin. Once the MTD is established, this portion of the study will close and the phase II will open to cohorts I and II at the recommended phase II dose (RP2D).
  Pembrolizumab: In this dose-finding cohort, pembrolizumab (MK-3475) were administered (cisplatin-eligible patients only) at starting dose 200mg IV every 21 days for 4 cycles to determine RP2D. Once MTD is established in phase Ib, pembrolizumab will be administered on phase II cohorts I and II at RP2D every 21 days for 5 cycles.
  Gemcitabine: For cisplatin-eligible patients on phase Ib, gemcitabine 1000mg/m2 IV, D1 and D8 every 21 days for 4 cycles.
  Cisplatin: For cisplatin-eligible patients, cisplatin 70mg/m2 IV will be administered D1 every 21 days for 4 cycles.
- Phase II Cohort I: Cisplatin Eligible- Pembrolizumab 200 mg: Cisplatin-eligible subjects receive gemcitabine/cisplatin every 21 days, repeated for 4 cycles. (Subjects with Ccr of 50-59 mL/min must follow split dosing of cisplatin over two days) . Pembrolizumab at RP2D is given every 21 days for 5 doses starting C1D8. Note: the last dose of pembrolizumab falls on what would be day 8 of a 5th 'chemo' cycle, however gemcitabine/cisplatin is NOT GIVEN. Subjects will then have consolidative surgery to remove their primary tumor within 2-7 weeks after their last dose of neoadjuvant therapy.
  Pembrolizumab: Once MTD is established in phase Ib, pembrolizumab will be administered on phase II cohorts I and II at RP2D every 21 days for 5 cycles.
  Gemcitabine: For cisplatin-eligible patients on phase II cohort 1, gemcitabine 1000mg/m2 IV, D1 and D8 every 21 days for 4 cycles.
  Cisplatin: For cisplatin-eligible patients, cisplatin 70mg/m2 IV will be administered D1 every 21 days for 4 cycles.
- Phase II Cohort II: Cisplatin Ineligible -Pembrolizumab 200 mg: Cisplatin ineligible (receive treatment in Phase II only): Cisplatin ineligible subjects receive gemcitabine every week (weekly) for three consecutive weeks, repeated every 28 days for 3 cycles. Pembrolizumab is given every 3 weeks for 5 doses starting with Cycle 1 Day 8 (C1D8). NOTE: due to the timing of gemcitabine cycles every 4 weeks, and every three week dosing of pembrolizumab, there are two doses of pembrolizumab given during cycle 2: days 1 and 22. Additionally, the last dose of pembrolizumab falls on what would be day 8 of a 4th 'chemo' cycle; however gemcitabine is NOT GIVEN.
Arm/Group | Phase 1b Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg | Phase II Cohort I: Cisplatin Eligible- Pembrolizumab 200 mg | Phase II Cohort II: Cisplatin Ineligible -Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 1/6 | 11/37 | 16/38
Serious Adverse Events (participants affected / at risk) | 1/6 | 17/37 | 17/38
Other Adverse Events (participants affected / at risk) | 6/6 | 37/37 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg (N=6) | Phase II Cohort I: Cisplatin Eligible- Pembrolizumab 200 mg (N=37) | Phase II Cohort II: Cisplatin Ineligible -Pembrolizumab 200 mg (N=38)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (2) | 1 (1) | 2 (2)
FEVER (General disorders) | 1 (1) | 1 (1) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CONFUSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
CREATININE INCREASED (Investigations) | 0 (0) | 1 (3) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
JEJUNAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
MOBITZ TYPE I (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 3 (4)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HEART FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort I: Cisplatin Eligible - Pembrolizumab 200 mg (N=6) | Phase II Cohort I: Cisplatin Eligible- Pembrolizumab 200 mg (N=37) | Phase II Cohort II: Cisplatin Ineligible -Pembrolizumab 200 mg (N=38)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 3 (3) | 5 (9)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 4 (5) | 11 (24)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 14 (17) | 6 (7)
ANEMIA (Blood and lymphatic system disorders) | 5 (14) | 23 (97) | 31 (112)
ANOREXIA (Metabolism and nutrition disorders) | 3 (5) | 16 (27) | 19 (32)
ANXIETY (Psychiatric disorders) | 1 (1) | 3 (5) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 3 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2) | 0 (0) | 12 (20)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 8 (9)
BLOATING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
BLURRED VISION (Eye disorders) | 3 (4) | 2 (2) | 3 (3)
BRUISING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 3 (7) | 19 (29) | 20 (28)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (10) | 16 (18)
CREATININE INCREASED (Investigations) | 2 (3) | 8 (18) | 8 (12)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 5 (6)
DEPRESSION (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 3 (5) | 7 (9) | 8 (13)
DIZZINESS (Nervous system disorders) | 3 (6) | 4 (4) | 8 (8)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 10 (10) | 1 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 9 (9) | 18 (34)
EDEMA LIMBS (General disorders) | 2 (3) | 9 (9) | 17 (23)
FATIGUE (General disorders) | 5 (13) | 30 (50) | 29 (48)
FEVER (General disorders) | 1 (1) | 4 (4) | 10 (13)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1) | 5 (9) | 1 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 6 (6)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1) | 3 (3) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 2 (6) | 5 (9) | 7 (14)
HYPERTENSION (Vascular disorders) | 4 (9) | 13 (25) | 18 (37)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (6) | 2 (3) | 10 (19)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 3 (6)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2) | 7 (8) | 3 (13)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (4) | 7 (10) | 6 (11)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
INSOMNIA (Psychiatric disorders) | 3 (3) | 5 (5) | 3 (3)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (3) | 3 (10) | 8 (24)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 3 (7) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 6 (10) | 21 (40) | 17 (27)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (7) | 18 (32) | 13 (26)
PAIN (General disorders) | 3 (3) | 5 (9) | 8 (13)
PALMAR-PLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 (7) | 9 (11) | 6 (7)
PLATELET COUNT DECREASED (Investigations) | 2 (4) | 15 (36) | 17 (39)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (3) | 8 (10) | 8 (9)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 (5) | 11 (14) | 7 (9)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1) | 4 (4) | 3 (4)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 3 (6) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (3) | 5 (6) | 8 (10)
SKIN INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
TINNITUS (Ear and labyrinth disorders) | 3 (5) | 5 (7) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (3) | 5 (5) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3) | 9 (13) | 12 (13)
URINARY TRACT PAIN (Renal and urinary disorders) | 1 (1) | 4 (5) | 3 (3)
VOMITING (Gastrointestinal disorders) | 2 (3) | 11 (14) | 8 (11)
WEIGHT LOSS (Investigations) | 3 (4) | 8 (11) | 4 (4)
WHITE BLOOD CELL DECREASED (Investigations) | 3 (7) | 7 (16) | 9 (24)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 2 (2) | 7 (8)
BLADDER INFECTION (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
BLADDER SPASM (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 2 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
BRONCHIAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
CHOLESTEROL HIGH (Investigations) | 0 (0) | 3 (3) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (4)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
EDEMA FACE (General disorders) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 0 (0) | 1 (1) | 2 (2)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
FLU LIKE SYMPTOMS (General disorders) | 0 (0) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 1 (1) | 3 (3)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 0 (0) | 3 (3) | 1 (1)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 6 (6) | 11 (15)
HEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HEMATURIA (Renal and urinary disorders) | 0 (0) | 5 (5) | 6 (8)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HOT FLASHES (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 4 (9)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 5 (12)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 5 (5) | 3 (3)
ILEAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 0 (0) | 5 (6) | 10 (15)
INFUSION RELATED REACTION (General disorders) | 0 (0) | 2 (2) | 0 (0)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE REACTION (General disorders) | 0 (0) | 1 (1) | 0 (0)
INJURY TO SUPERIOR VENA CAVA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LOCALIZED EDEMA (General disorders) | 0 (0) | 3 (3) | 2 (2)
MUCOSITIS ORAL (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (7)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (9) | 7 (8)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
PANCREATIC ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 4 (5) | 4 (7)
PENILE PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PHLEBITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (12) | 3 (3)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
RHINITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
SCROTAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 0 (0) | 5 (5) | 2 (3)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 (0) | 5 (6) | 3 (3)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
WATERING EYES (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
WEIGHT GAIN (Investigations) | 0 (0) | 2 (2) | 2 (2)
AKATHISIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CHILLS (General disorders) | 0 (0) | 0 (0) | 4 (4)
CONFUSION (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
HEART FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4)
HYPERURICEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
LYMPHEDEMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 0 (0) | 2 (2)
MUCOSAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
NAIL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 2 (3)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PHARYNGEAL MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
SCROTAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VAGINAL PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02365766/Prot_SAP_000.pdf